CLINICAL TRIAL: NCT06694831
Title: Evaluation of Anxiety of Patients Coming to Our Country for Bariatric Surgery Through Health Tourism Using Psychiatric Tests
Brief Title: Health Tourism in Bariatric Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: İlke Dolgun (Other)
Responsible Party: Sponsor-Investigator, İlke Dolgun, Assoc. prof, Istinye University
Organization: Istinye University (Other)
Other Study IDs: hakan health tourism
Record Dates: First submitted 2024-10-21; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to examine whether patients who come to our country for bariatric surgery via health tourism have any concerns during this process, and if they do, to determine the level of their concerns through psychometric tests, to determine the reasons for their concerns (is it related to travel, going to another country, hospital, surgery, etc.) and whether their concerns decrease after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who came to our country through health tourism
* Patients with indications for bariatric surgery
* Patients over the age of 18

Exclusion Criteria:

* Patients under 18 years of age
* Patients with psychiatric, neurological diseases or mental retardation that prevent them from completing psychometric tests
* Patients with bariatric surgery indications other than health tourism
* Patients who do not agree to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients over the age of 18 who came to our country for bariatric surgery through health tourism
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2025-01-25 (Estimated); Study Completion 2025-02-25 (Estimated)

PRIMARY OUTCOMES:
anxiety scale | 1 month
  to examine whether they have concerns

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye Üniversity, Istanbul, Merkez Mahallesi, Turkey (Türkiye)

REFERENCES:
- [Result] Zuberi S, Egiz A, Iqbal H, Jambulingam P, Whitelaw D, Adil T, Jain V, Al-Taan O, Munasinghe A, Askari A, Aly MK, Iqbal FM. Characterizing barriers and facilitators of metabolic bariatric surgery tourism: a systematic review. Br J Surg. 2024 Mar 2;111(3):znae060. doi: 10.1093/bjs/znae060. PMID 38547416
- [Result] Demir Y, Özpınar S. Evaluation of the Effect of Body Image Perception on Patient Satisfaction and Quality of Life in Medical Tourists Undergoing Bariatric Metabolic Surgery. Int Journal Of Health Manag. And Tourism 2024, 9(1), 62-75.